CLINICAL TRIAL: NCT04658381
Title: Genetic Analysis and Multimodal Retinal Imaging of Asymptomatic Fovea Plana Cases in the General Population
Acronym: APOGEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RLX_2020_27
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2024-01

CONDITIONS: Fovea Plana; Albinism
Keywords: Carriers; General population
MeSH Terms: conditions — Albinism | interventions — Genetic Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genetic analysis (Experimental)
  Interventions: Genetic: Genetic analysis; Procedure: Ophthalmologic exam

INTERVENTIONS:
Genetic: Genetic analysis — Patient exome sequencing will be performed by Illumina technology on the NextSeq 550 sequencer. Briefly, the exons of the genes are selected by capture and are amplified by PCR simultaneously, in a single reaction, and then sequenced by Illumina technology. The analysis will only concern genes involved in albinism and in genetic pathologies associated with fovea plana.
Procedure: Ophthalmologic exam — Standard ophthalmologic assessment (measurement of visual acuity, measurement of intraocular pressure, slit lamp examination), OCT-B scan, OCT-Angiography, Adaptive optics

SUMMARY:
Albinism is a genetic condition, resulting from mutations in at least 19 known genes responsible for the production of melanin in the skin, hair and eyes.

Ophthalmological manifestations are a constant feature of this disease. Albinism is believed to be responsible for 5% of visual impairments worldwide and all albino patients have some degree of fovea plana. In the milder forms, it is a slightly less marked foveolar depression with conservation of the normal diameter of the cones and, therefore, good visual function.

In addition to its known association with various ocular pathologies such as albinism, aniridia, nanophthalmia and retinopathy of prematurity, fovea plana was found in 3% of a population of normal children (without known ocular or systemic pathology) in a study conducted in 2014 to determine a pediatric normative basis for macular volume measured by optical coherence imaging (Stratus OCT).

More recently, a study carried out at the Hospital Foundation Adolphe de Rothschild showed that at least 35% of parents of albino children, who are totally asymptomatic, present with fovea plana in OCT. This frequency is higher than the 3% prevalence of fovea plana in asymptomatic subjects without a family history of albinism, suggesting a modulation of heterozygosity for a known gene for albinism.

The aim of this study is to verify, in patients with fortuitously discovered fovea plana (preoperative OCT for cataract surgery), with conservation of visual function and without known or manifest albinism, whether they are carriers of mutation in one of the genes referenced for albinism. This will also allow us to characterize these foveolar profiles in OCT according to the classification of Thomas et al., as well as in terms of retinal capillary density in OCT-Angiography, in order to know whether it is the same type of fovea plana or if the phenotype differs depending on the genetic damage.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old;
* Diagnosis of fovea plana in one or both eyes, confirmed by two ophthalmologists blinded to each other from OCT-B imaging;

Exclusion Criteria:

* Known Albinism
* Known family history of albinism
* History of eye surgery other than cataract
* Alteration of macular visual function (loss of visual acuity independent of a disorder of the environments, central scotoma, metamorphopsies, etc.)
* Presence of another anomaly in OCT in addition to the fovea plana (epiretinal membrane, damage to the external retina, etc.)
* Syndromic fovea plana
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Describe the results of genetic analysis for the various variants of known genes involved in albinism and in genetic pathologies associated with fovea plana | 2 years
  Genetic sampling carried out for the study. Patient exome sequencing. The analysis will only concern genes involved in albinism and in genetic pathologies associated with fovea plana

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël LEJOYEUX, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, France

REFERENCES:
- [Result] Lejoyeux R, Michaud V, Le Boite H, Plaisant C, Helot I, Philippe E, Lasseaux E, Vasseur V, Fessard K, Picard H, Le Cossec C, Bruneau S, Le Mer Y, Arveiler B, Couturier A, Bonnin S. Genetic analysis of participants with foveal hypoplasia. Ophthalmic Genet. 2025 Dec;46(6):559-562. doi: 10.1080/13816810.2025.2520411. Epub 2025 Jun 23. PMID 40546025